CLINICAL TRIAL: NCT07186543
Title: Co-Designing a Virtual Reality Intervention to Enhance Skill Development With Adolescents Hospitalized for Suicide-Related Crises
Brief Title: Co-Designing a Virtual Reality Intervention to Enhance Skill Development
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: MQ Mental Health Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-0388
Record Dates: First submitted 2025-09-11; First posted 2025-09-22 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Suicide
MeSH Terms: conditions — Suicide | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Control (Active Comparator): Cognitive Behavioral Therapy (CBT) Worksheets
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT) Worksheets
- PrESR Intervention (Experimental): Cognitive Behavioral Therapy (CBT) Worksheets; Virtual Reality (VR) Enhanced CBT Skill/Practice; Safety Planning
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT) Worksheets; Behavioral: Practice Experiences for School Reintegration (PrESR)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) Worksheets — The researchers will provide instructions for participants to complete a packet of worksheets teaching introduction to cognitive behavioral therapy (CBT), affect regulation, cognitive restructuring, and problem solving.
Behavioral: Practice Experiences for School Reintegration (PrESR) — Participants will receive an overview of cognitive behavioral therapy skills in virtual reality (VR) and then have the opportunity to practice using skills in a brief immersive experience designed to mimic difficult school and social experiences. Session begin with goal setting and conclude with a debrief summary following the VR experience. Prior to discharge and following the conclusion of the VR sessions, participants will be invited to collaborate on a safety planning intervention informed by their experiences in VR that addresses school and social experiences.
  Arms: PrESR Intervention

SUMMARY:
This study is refining and pilot testing a novel Virtual Reality (VR) supplement for inpatient treatment: the Practice Experiences for School Reintegration (PrESR) program. The PrESR provides immersive school and social experiences for inpatient adolescents (with suicidal-related admissions) to practice skills in real-world settings with the guidance of a trained clinician within the confines of a hospital. The initial intervention was based on feedback from adolescent hospitalized for suicide-related crises, and school and hospital professionals, but did not provide tailored experiences to address the individual needs of ethnic-racial, gender, and sexual minoritized adolescents. Therefore, the VR environment of PrESR was adapted based on input from adolescents with previous suicide-related crises identifying as ethnic, racial, sex, or gender minoritized. This pilot randomized controlled trial (RCT) aims to explore the feasibility, acceptability, and facilitators/barriers to implementation of the adapted version of PrESR for improving outcomes in hospitalized adolescents. This study is not powered to test hypotheses; however, in addition to assessing feasibility, acceptability, and barriers/facilitators, this pilot trial will assess candidate intermediary and outcome measures.

DETAILED DESCRIPTION:
This study recruits a prospective sample of youth hospitalized for suicide-related crises. Target sample size is approximately N = 26 enrolled adolescents, with the intention of recruiting at least 16 participants who identify as ethnic, racial, sex, or gender minoritized. The pilot RCT includes two conditions: an enhanced treatment as usual condition and an experimental condition. All participants will receive standard treatment, as well as researcher provided worksheets addressing introduction to cognitive behavioral therapy, cognitive restructuring, problem-solving, and affect regulation. Participants randomized to the experimental condition will also receive one or more sessions with PrESR. Outcomes will be assessed during hospitalization and again 3-weeks following hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Current hospitalization for suicidal thoughts and behaviors
* Ages 13-18
* Clinician approval
* Ability to speak, read, and understand English sufficiently to complete study procedures
* Consent of a parent/legal guardian (in English or Spanish; for minor participants)
* Adolescent assent or consent (in English)

Exclusion Criteria:

* Evidence of active psychosis
* Evidence of intellectual disability
* Risk for cybersickness (greater or equal to 50th percentile as measured on the Motion Sickness Susceptibility Questionnaire).

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients in the Target Population Who Agree to Participate | Baseline
  Recruitment rate determined based on the proportion of adolescents providing assent and parents or legal guardians providing permission relative to the number of parents or legal guardians approached.
Proportion of Patients in the Target Population Excluded Due to Motion Sickness Screening | Baseline
  Rate of recruitment related to motion sickness determined based on the proportion of assented adolescents whose scores were >/= than 50th percentile on motion sickness questionnaire relative to the number of assented adolescents.
Proportion of Participants Who Complete All Study Procedures | up to 3-weeks following hospital discharge
  Proportion of participants who complete all study procedures determined based on the proportion of adolescents completing study procedures at Baseline and 3-week follow-up relative to the total number of adolescents participating in that condition.
Average Number of Hours to Complete Assessments at Each Time Point | up to 3-weeks following hospital discharge
  Time to complete assessments, assessments are expected to last less than 4 hours.
Average Number of Minutes to Complete Each Intervention Session | Baseline
  Time to complete intervention sessions, each session is expected to last less than 60 minutes. Average calculated by summing all sessions in each condition and dividing by total number of sessions.
Percentage of Adolescent Participants in Which Intervention Delivered With Greater Than or Equal to 80% Fidelity | Baseline
  Percentage of participants in which adherence to delivery of key components of intervention (i.e., skill lessons or practice sessions) across sessions in each condition was 80% or greater. Adherence calculated based on the number of key components completed relative to the total number of key components expected to be completed for each participant.
Percentage of Adolescent Participants With Average Acceptability Scores Less Than or Equal to 2 | Baseline
  Percent of adolescents with average acceptability score less than or equal to 2 (or "agree") on a structured feedback form developed by the researchers. The structured feedback form includes an average of four items related to acceptability on a five-point scale from 1 (strongly agree) to 5 (strongly disagree), with lower scores reflecting higher acceptability.
Adolescents' Perceptions of Acceptability | Baseline
  Qualitative feedback provided by adolescents receiving the intervention about acceptability of the intervention, with the two most common points of feedback collected from a structured interview reported.

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Marraccini, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Adolescent Psychiatry Inpatient Unit, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC